CLINICAL TRIAL: NCT04388501
Title: A Single-center, Open-label, Randomized, Three-way Cross-over Study Evaluating Drug Drug Interaction Between JNJ-70033093 and Atorvastatin in Healthy Participants
Brief Title: A Study Evaluating Drug Drug Interaction Between Milvexian and Atorvastatin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108776; 2019-004640-29 (EudraCT Number); 70033093THR1002 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — milvexian; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence ABC (Experimental): Participants will receive milvexian capsule once daily (qd) for 5 days (Treatment A) in Period 1 followed by Atorvastatin tablets qd for 5 days (Treatment B) in Period 2 followed by milvexian capsules qd and atorvastatin tablets qd for 5 days (Treatment C) in Period 3. Each period is separated by a washout period of 7 days.
  Interventions: Drug: Milvexian; Drug: Atorvastatin
- Treatment Sequence BCA (Experimental): Participants will receive Treatment B in Period 1 followed by Treatment C in Period 2 and Treatment A in Period 3. Each Period is separated by a washout period of 7 days.
  Interventions: Drug: Milvexian; Drug: Atorvastatin
- Treatment Sequence CAB (Experimental): Participants will receive Treatment C in Period 1 followed by Treatment A in Period 2 and Treatment B in Period 3. Each Period is separated by a washout period of 7 days.
  Interventions: Drug: Milvexian; Drug: Atorvastatin
- Treatment Sequence CBA (Experimental): Participants will receive Treatment C in Period 1 followed by Treatment B in Period 2 and Treatment A in Period 3. Each Period is separated by a washout period of 7 days.
  Interventions: Drug: Milvexian; Drug: Atorvastatin
- Treatment Sequence ACB (Experimental): Participants will receive Treatment A in Period 1 followed by Treatment C in Period 2 and Treatment B in Period 3. Each Period is separated by a washout period of 7 days.
  Interventions: Drug: Milvexian; Drug: Atorvastatin
- Treatment Sequence BAC (Experimental): Participants will receive Treatment B in Period 1 followed by Treatment A in Period 2 and Treatment C in Period 3. Each Period is separated by a washout period of 7 days.
  Interventions: Drug: Milvexian; Drug: Atorvastatin

INTERVENTIONS:
Drug: Milvexian — Participants will receive milvexian capsules orally qd for 5 days as per the assigned treatment sequence.
  Other Names: BMS-986177, JNJ-70033093
Drug: Atorvastatin — Participants will receive atorvastatin tablets orally qd for 5 days as per the assigned treatment sequence.

SUMMARY:
The purpose of this study is to evaluate the potential pharmacokinetics (PK) interaction between milvexian and atorvastatin (and its metabolites) in healthy participants at steady state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, Electrocardiogram (ECG), and laboratory test results, including serum chemistry, blood coagulation, hematology, and urinalysis, performed at screening.
* Normal renal function at screening as evidenced by an estimated glomerular filtration rate (eGFR) of greater than or equal to (>=) 90 milliliter per minute per 1.73 square meters (mL/min/1.73 m^2) calculated with the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
* Must sign an informed consent form (ICF) indicating they understand the purpose of, and procedures required for, the study and are willing to participate in the study
* If a woman, except for postmenopausal women, must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and urine (beta-hCG) pregnancy test on Day 1 of each treatment period
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies

Exclusion Criteria:

* Participant is a woman who is pregnant, breastfeeding, or planning to become pregnant during this study or within 34 days after the last study drug administration
* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, gastrointestinal disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, coagulation, clinical chemistry (including thyroid-stimulating hormone [TSH] at screening only), or urinalysis at screening or on Day 1 prior to the first dosing, including: Hemoglobin and hematocrit less than (<) lower limit of normal; Platelet count < lower limit of normal; and activated partial thromboplastin time (aPTT) or prothrombin time (PT) greater than (>) 1.2* upper limit of normal (ULN)
* Clinically significant abnormal physical examination, vital signs, or 12 lead ECG at screening or at admission to the study center on Day 1 prior to first dosing, as deemed appropriate by the investigator
* Participants with a history of excessive menstrual bleeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Milvexian at Steady State | Predose, 0.5, 1, 2, 3, 4, 6, 10, 12, 14 hours after drug administration on Day 5 in Period 1, 2, 3
  Cmax is the maximum observed plasma concentration of milvexian at Steady State.
Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24hours]) of Milvexian at Steady State | Predose, 0.5, 1, 2, 3, 4, 6, 10, 12, 14 hours after drug administration on Day 5 in Period 1, 2 and 3
  AUC(0-24 hours) is the area under the plasma concentration-time curve from time zero to 24 hours of milvexian at Steady State.
Maximum Observed Plasma Concentration (Cmax) of Atorvastatin at Steady State | Predose, 0.5, 1, 2, 3, 4, 6, 10, 12, 14 hours after drug administration on Day 5 in Period 1, 2, 3
  Cmax is the maximum observed plasma concentration of Atorvastatin at Steady State.
Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24hours]) of Atorvastatin in Healthy Participants at Steady State | Predose, 0.5, 1, 2, 3, 4, 6, 10, 12, 14 hours after drug administration on Day 5 in Period 1, 2 and 3
  AUC(0-24 hours) is the area under the plasma concentration-time curve from time zero to 24 hours of Atorvastatin at Steady State.

SECONDARY OUTCOMES:
Cmax of Milvexian After a Single Dose Administration | Predose, 0.5, 1, 2, 3, 4, 6, 10, 12, 14, 24, 48, 72 hours after drug administration on Day 1 in Period 1, 2, 3
  Cmax is the maximum observed plasma concentration of milvexian after single dose administration on Day 1.
AUC(0-24 hours) of Milvexian After a Single Dose Administration | Predose, 0.5, 1, 2, 3, 4, 6, 10, 12, 14, 24 hours after drug administration on Day 1 in Period 1, 2, 3
  AUC(0-24 hours) is the area under the plasma concentration-time curve from time zero to 24 hours of milvexian after single dose administration on Day 1.
Cmax of Atorvastatin After a Single Dose Administration | Predose, 0.5, 1, 2, 3, 4, 6, 10, 12, 14, 24, 48, 72 hours after drug administration on Day 1 in Period 1, 2, 3
  Cmax is the maximum observed plasma concentration of Atorvastatin after single dose administration on Day 1.
AUC(0-24 hours) of Atorvastatin After a Single Dose Administration | Predose, 0.5, 1, 2, 3, 4, 6, 10, 12, 14, 24 hours after drug administration on Day 1 in Period 1, 2, 3
  AUC(0-24 hours) is the area under the plasma concentration-time curve from time zero to 24 hours of Atorvastatin after single dose administration on Day 1.
Number of Participants with Adverse Event as a Measure of Safety and Tolerability | Up to 3.4 months
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Change From Baseline in Activated Partial Thromboplastin Time (aPTT) | Baseline, Day 2 and Day 6
  Activated partial thromboplastin time measures the time to clot formation via the intrinsic (contact) and common pathways, and is dependent on activation of contact factors (such as FXI). The assay is triggered in citrated platelet-poor plasma by addition of phospholipids, a contact activator (typically a negatively charged substance, as kaolin or ellagic acid), and calcium. The time taken for a fibrin clot to form is measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency